CLINICAL TRIAL: NCT02339714
Title: Effect Comparison of Acupuncture Combined With Moxibustion and Loratadine for Perennial Allergic Rhinitis: a Randomized Controlled Trial
Brief Title: Effectivness and Safety of Acupuncture Combined With Moxibustion for Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhao Hong (Other)
Collaborators: China Academy of Chinese Medical Sciences (Other); Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, Zhao Hong, Vice president of acupuncture and moxibustion hospital, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAMH001
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: allergic rhinitis; acupuncture; moxibustion; efficacy; safety
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — Loratadine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture combined moxibustion (Experimental): Acupuncture at Hegu(LI4),Yingxiang(LI20),Chize(LU5),Sibai(ST2), Yintang(EX-HN3),Shangyingxiang(EX-HN8),Shangxing(GV23),Dazhui(Du14). Needle warming moxibustion at Dazhui(Du14). Patients will be treated once per day for 30 min, 3 times in a weeks for 4 weeks.
  Interventions: Other: acupuncture combined moxibustion
- loratadine (Active Comparator): Loratadine taken orally, 10mg/day in the morning
  Interventions: Drug: Loratadine

INTERVENTIONS:
Other: acupuncture combined moxibustion — Points: Hegu(LI4),Yingxiang(LI20),Chize(LU5),Sibai(ST2), Yintang(EX-HN3),Shangyingxiang(EX-HN8),Shangxing(GV23),Dazhui(Du14).
  Pierced the skin, needles are inserted 0.5 to 2cm into the acupoints. Each needle are roated until the participants and the practitioner felt de-qi sensation. After that, moxibustion is applied to Dazhui(Du14). A 1cm long moxa cone is putted on the top of the needle at the acupoint, then ignite moxa cone until the cone is burn. The needles are left in place for 30 minutes. once every two days, 3 times in a week for consecutive 4 weeks, 12 times altogether.
  Other Names: warming needle
  Arms: Acupuncture combined moxibustion
Drug: Loratadine — Loratadine will be taken orally at the dose of 10mg/day in the morning. Each treatment cycle will be given for continuous 4 weeks.
  Arms: loratadine

SUMMARY:
A multi-centre clinical trial done by us（ISRCEN90807007）showed that active acupuncture had significantly greater effect on symptoms of allergic rhinitis than either sham acupuncture or no active treatment. The object of that study was to evaluate the effectiveness and safety of acupuncture for allergic rhinitis. As an explanatory research, acupuncture was defined as the only intervention for treatment group and sham acupuncture, no active treatment as its control groups. Besides, acupuncture combined moxibustion showed better and longer effect than acupuncture on allergic rhinitis patients in our previous pilot study. According to this result, we are taking a pragmatic randomized controlled trial to further evaluate whether acupuncture combined moxibustion is more effective than conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

Each participant must have a diagnosis of AR by an otolaryngology doctor, according to the criteria listed in "Allergic Rhinitis and its Impact on Asthma" (ARIA 2008) Symptoms that had persisted for more than 4 days per week for more than four consecutive weeks.

At least one of the following rhinitis-associated conditions: nasal obstruction, rhinorrhea, sneezing and nasal itching.

At least one positive result on an allergy skin prick reaction test at screening.

-

Exclusion Criteria:

Active tuberculosis Autoimmune disorders Severe chronic inflammatory diseases History of anaphylactic reactions Specific immunotherapy >3 years Simultaneous participation in other clinical trials Serious acute or chronic organic disease or mental disorder Congenital nasal abnormalities Pregnancy or breast feeding Blood coagulation disorder and/or current use of anticoagulants Allergy desensitisation therapy (current, during the past two years, or planned in the next two years) Previous systemically administered corticosteroids, antihistamines, or decongestants in the last 1 months prior to enrollment

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly average of the participants' total nasal symptom score (TNSS) at the 4th week. | at the 4th week

SECONDARY OUTCOMES:
Change from baseline in the weekly average of the participants' total non-nasal symptom score (TNNSS) at the 4th week | at the 4th week
Change from baseline in Quality of life questionnaire (QLQ) at the 4th week | at the 4th Week

CONTACTS AND LOCATIONS:
Overall Officials: Liu Baoyan, Master, Principal Investigator — Vice President of China Academy of Chinese Medical Sciences
Locations (3):
- China (3):
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Institute of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Mentougou Hospital of TCM, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Sun Y, Zhao H, Ye Y, Nie W, Bai W, Liu J, Li S, Wang F, Han M, He L. Efficacy and safety of using a warming needle for persistent allergic rhinitis: study protocol for a randomized controlled trial. Trials. 2016 Jun 30;17(1):305. doi: 10.1186/s13063-016-1432-z. PMID 27363578